CLINICAL TRIAL: NCT02238613
Title: Intraluminal Implantation of Radioactive Stents for Treatment of Unresectable Biliary Tract Cancer
Brief Title: Radioactive Stents for Treatment of Unresectable Biliary Tract Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: 307 Hospital of PLA (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Changhai Hospital (Other)
Responsible Party: Principal Investigator, yan liu, PhD, MD. Chairman of Department of Gastroenterology and Hepatology, 307 Hospital of PLA, 307 Hospital of PLA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: yanliu307; 307xhk (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2014-08-25; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Intrahepatic Cholangiocarcinoma; Cholangiocarcinoma of the Extrahepatic Bile Duct; Ampullary Carcinoma; Biliary Obstruction
Keywords: Radioactive stents; Brachytherapy; Biliary obstruction; Intrahepatic Cholangiocarcinoma; Cholangiocarcinoma of the Extrahepatic Bile Duct; ampullary carcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- radioactive stent (Experimental): The radioactive stent carrying seeds iodine 125 is made of Polytetrafluoroethylene. It will be implanted in the common bile duct by ERCP(endoscopic retrograde cholangiopancreatography) of the irradiation group patients.
  Interventions: Device: radioactive stent
- plastic stent (Other): The plastic stent is made of polyethylene. It will be implanted in the common bile duct by ERCP(endoscopic retrograde cholangiopancreatography) of the conventional group patients.
  Interventions: Device: plastic stent

INTERVENTIONS:
Device: radioactive stent — radioactive stent carrying seed iodine 125
  Other Names: brand names: carriable radioactive bile duct plastic stent; serial numbers and code name: PBS1-A/B-10/160/140
  Arms: radioactive stent
Device: plastic stent — common plastic stent without carrying seed iodine 125
  Arms: plastic stent

SUMMARY:
The purpose of this study is to determine whether radioactive stents and common used plastic stents are effective and safety in the treatment of unresectable biliary tract cancer.

DETAILED DESCRIPTION:
Patients with unresectable biliary tract cancer (intrahepatic or extrahepatic cholangiocarcinoma, or ampullary carcinoma) were enrolled and placed with a stent loaded with radioactive seeds (irradiation stent group) or a conventional plastic stent (traditional stent group). After stent placement, the outcomes were compared in terms of tumor response, progression-free survival, overall survival time, and complications related to the procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible if they had received a histopathological or cytologic diagnosis of nonresectable, recurrent, or metastatic biliary tract carcinoma (intrahepatic or extrahepatic cholangiocarcinoma,or ampullary carcinoma)
* Patients aged between 18 and 80 years
* an estimated life expectancy of more than 3 months
* Disease had to be measurable by computed tomography scan (as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.0 criteria
* TNM stage III-IV
* no evidence of cancer of another organ.
* no prior chemotherapy for advanced disease was allowed, but adjuvant/neoadjuvant therapy was allowed
* Karnofsky index of ≥60%
* ECOG index ≥2
* previous technically successful stenting or ENBD derange
* Accept of informed consent

Exclusion Criteria:

* Clinically significant cardiovascular disease
* coagulation disorders
* contraindication of Endoscopic
* pregnant or breastfeeding women
* known sensitivity sensitivity to investigated agents or components
* recent invasive procedure
* prior chemotherapy or radiotherapy for biliary cancer
* refusal of informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Tumor Response rate | 3 months
  The investigators will conduct CT test or MRI scan after the implantation of the stents in order to measure the tumor size of each patients and evaluate the best tumor response according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.0).

SECONDARY OUTCOMES:
Progression-free survival | 6 months
  In order to research the progression-free survival, the investigators will check the presence of progression disease for each patients until the date of disease progression or death.
overall survival | follow-up in interval of stent insertion and death (1 years)
  Overall survival was calculated from the date of randomization until the date of death.
Adverse events | 1 year
  Individual adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, Doctor, Principal Investigator — 307 hospital of PLA, Beijing, China
Locations (1):
- 307 hospital of PLA, Beijing, Beijing Municipality, China